CLINICAL TRIAL: NCT02268565
Title: Preventing the Inflammatory Response to Experimentally-induced Insomnia Symptoms
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Monika Haack, Assistant Professor of Neurology, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2014P000269
Record Dates: First submitted 2014-09-23; First posted 2014-10-20 (Estimated); Last update posted 2017-03-15 (Actual); Status verified 2017-03

CONDITIONS: Insomnia
Keywords: sleep, insomnia, inflammation, pain; Insomnia symptom induction/placebo; Insomnia symptom induction/aspirin
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Inflammation; Pain | interventions — Aspirin; Anti-Inflammatory Agents, Non-Steroidal

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Insomnia symptom induction/placebo (Placebo Comparator): Daily intake of pill at bedtime over 2-week period prior to and during the 5-day in-hospital stay
  Interventions: Drug: Placebo
- Insomnia symptom induction/aspirin (Experimental): Daily intake of pill at bedtime over 2-week period prior to and during the 5-day in-hospital stay
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: Aspirin — 81mg aspirin daily at bedtime over a 2 week period
  Other Names: non-steroidal anti-inflammatory drug
  Arms: Insomnia symptom induction/aspirin
Drug: Placebo — pill that looks like aspirin without the effects of aspirin
  Arms: Insomnia symptom induction/placebo

SUMMARY:
The main purpose of this study is to learn about the effects of sleep disruption (two days in a row where sleep is shortened and disrupted) on inflammation, mood (how you feel), and pain processing (your own experiences/perceptions of pain). In this research project, we are trying to figure out if we can change the effects of sleep disruption on inflammation, mood, and pain. Therefore, we will study whether taking a low-dose aspirin pill every day over 2 weeks can change how we respond to sleep disruption. For example, does the sensitivity to pain (e.g., how intense the feeling of pain is if we put our hand in very hot or very cold water) change with sleep disruption, and can low-dose aspirin influence this change. We are also interested in seeing how inflammation changes in relation to your own perceived experience of pain.

DETAILED DESCRIPTION:
Sleep that is deficient in quantity or quality leads to upregulation of inflammatory markers (Mullington et al., 2010). In particular, interleukin (IL)-6 and prostaglandin (PG) E2 are elevated in experimental models of sleep restriction or total sleep deprivation, as well as in insomnia. Inflammation is thought to be a key mechanism through which insufficient sleep increases the risk of developing or exacerbating various disorders, including cardiovascular and metabolic disorders (Mullington et al., 2009), as well as pain-related disorders (Haack et al., 2009c). With respect to pain, markers such as IL-6 and PGE2 are able to sensitize pain transmission neurons, thereby increasing their responsiveness to stimulation. In the context of insufficient sleep, both IL-6 and PGE2 have been shown to be associated with increased spontaneous pain (Haack et al., 2007;Haack et al., 2009a), suggesting their mediating role in pain amplification as a consequence of insufficient sleep.

These findings raise the question of whether pain amplification can be dampened by preventing the inflammatory increase in response to insufficient sleep.

The primary goal of this pilot project is to gather preliminary support for the hypothesis that deficient sleep leads to pain amplification through an inflammatory mechanism.

In addition to the primary goal of this proposal, the secondary goal is to gather preliminary data on the effects of aspirin on blood pressure regulation. Cardiovascular disease is the leading cause of death in the United States. A modest reduction of blood pressure (BP; i.e., 3 to 5 mmHg) in the population will produce a significant fall in serious cardiovascular events (Turnbull, 2003). It has been reported that low-dose aspirin may significantly reduce BP (i.e., 6 to 7 mmHg) when taken at bedtime (Hermida et al., 1994;Hermida et al., 1997;Hermida et al., 2003b;Hermida et al., 2003a;Hermida et al., 2005a;Hermida et al., 2005b). Aspirin, when taken at bedtime, may modulate 24h blood pressure by decreasing the nocturnal rise of renin-angiotensin-aldosterone system (RAAS) activity (Snoep et al., 2009) and attenuating the nocturnal drop in nitric oxide (NO) production (Hermida et al., 2005b). However, the underlying mechanisms are still unknown. Therefore, the second goal of this pilot project is to investigate the potential mechanisms contributing to BP reduction in response to aspirin taken at bedtime.

ELIGIBILITY:
Inclusion Criteria:

* Women and men between the ages 18-35 years
* Body mass index (BMI) between 18.5 and 30.0 kg/m2
* For female participants: regular menstrual cycles, no significant discomfort during pre-menses/menses
* Daily sleep duration between 7.0-9.0 hours, verified by sleep log/actigraphy data for two weeks
* Habitual sleep period must begin within one hour of 2300h (to ensure normal entrainment)
* Blood chemistry in the normal range

Exclusion Criteria:

* Active infection/disease.
* History of psychiatric, neurological, pain-related, immune, gastrointestinal, or cardiovascular disease; significant allergy; Raynaud's syndrome.
* History of intolerance or allergy to non-steroidal anti-inflammatory drugs (NSAID)
* Esophageal reflux; gastric or duodenal ulcers; or asthma
* Pregnant/nursing.
* Respiratory disturbance index of >5 events/hour on polysomnographic sleep study, periodic leg movement index (PLMI) >15/hour; sleep efficiency <80% (findings indicative of a sleep disorder).
* Regular medication use other than oral contraceptives.
* Donation of blood or platelets 3 month prior to or in-between in-hospital visits.
* Substance abuse.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2014-10; Primary Completion 2016-10 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Inflammation | Measured in plasma and urine 3 times/day over the 5-day in-hospital stay (after 2 weeks of pill admin)
  interleukin 6

SECONDARY OUTCOMES:
Pain sensitivity | Measured once per day during in-hospital days 1-5 (after 2 weeks of pill admin)
  Thermode will be attached to the skin and participant has to rate the intensity of the heat or cold sensation via visual analog scales

OTHER OUTCOMES:
Pain modulation | Measured once per day during in-hospital days 1-5
  Participant has to immerse foot into cold or hot water and rate the intensity of heat pain or cold stimuli applied to the arm on visual analog scales

CONTACTS AND LOCATIONS:
Overall Officials: Monika Haack, PhD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States